CLINICAL TRIAL: NCT02839629
Title: Long-term Epidemiological Follow-up of Non-small Cell Lung Cancer in Scandinavia
Acronym: SCAN-LEAF
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-319
Record Dates: First submitted 2016-07-12; First posted 2016-07-21 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort 1: National patient cohorts in Scandinavia: Scandinavian countries: Denmark, Norway and Sweden Cohort 1 will include all patients with a diagnosis of NSCLC between 2005 and 2013
- Cohort 2: Electronic Medical Records based cohort (Sweden): Patient as data is available (~2010) to 2013

SUMMARY:
A study to describe and evaluate patient characteristics and clinical outcomes in Subjects with diagnosed Non Small Lung Cell Cancer in Sweden, Norway and Denmark.

ELIGIBILITY:
Inclusion Criteria:

Patients with a histologically confirmed diagnosis of NSCLC (squamous, adenocarcinoma, not otherwise specified NSCLC [NSCLC NOS]) identified in the Cancer registers

Exclusion Criteria:

* Age under 18 years at time of diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 5657 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Overall survival based on Response Evaluation Criteria in Solid Tumors (RECIST) | Approximately 2 years
  Overall survival is defined as the time from start of treatment to the end of follow-up; Clinical outcomes will be assessed among NSCLC patients with advanced (stage IIIB and above) and earlier stage (stages I to IIIA) disease
Progression free survival based on Response Evaluation Criteria in Solid Tumors (RECIST) | Approximately 2 years
  Progression free survival is defined as the time from date of treatment start to either the first disease progression date or last known tumor assessment date or death; Clinical outcomes will be assessed among NSCLC patients with advanced (stage IIIB and above) and earlier stage (stages I to IIIA) disease
Time to progression based on Response Evaluation Criteria in Solid Tumors (RECIST) | Approximately 2 years
  Time to progression is defined as time from start of therapy until tumor progression; Clinical outcomes will be assessed among NSCLC patients with advanced (stage IIIB and above) and earlier stage (stages I to IIIA) disease
Disease control rate; defined as total number of patients whose Best Overall Response(BOR)= Complete Response(CR), Partial Response(PR) or Stable Disease(SD), divided by total number of patients | Approximately 2 years
  Clinical outcomes will be assessed among NSCLC patients with advanced (stage IIIB and above) and earlier stage (stages I to IIIA) disease; BOR: Best Overall Response, CR: Complete Response, PR: Partial Response, SD: Stable Disease
Partial Response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) | Approximately 2 years
  Partial response is defined as a record of at least a 30% decrease in the sum of diameters of target lesions, from the baseline sum; Clinical outcomes will be assessed among NSCLC patients with advanced (stage IIIB and above) and earlier stage (stages I to IIIA) disease
Complete response based on Response Evaluation Criteria in Solid Tumors (RECIST) | Approximately 2 years
  Complete response is defined as a record of disappearance of all target lesions; Clinical outcomes will be assessed among NSCLC patients with advanced (stage IIIB and above) and earlier stage (stages I to IIIA) disease
Percent of patients with an adverse event (AE) | Approximately 2 years
  Patients with advanced stage (stage IIIB and above) disease; AEs are defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Percent of patients with an adverse event (AE) | Approximately 2 years
  Patients with earlier stage (stages I to IIA) disease; AEs are defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product

SECONDARY OUTCOMES:
Body Mass Index (BMI) of NSCLC patients at diagnosis | At baseline visit
Smoking habits of NSCLC patients at diagnosis | At baseline visit
Age of NSCLC patients at diagnosis | At baseline visit
NSCLC clinical subtype of NSCLC patients at diagnosis | At baseline visit
Tumor node metastasis classification of NSCLC patients at diagnosis | At baseline visit
Charlson Comorbidity index of NSCLC patients at diagnosis | At baseline visit
Drug utilization after NSCLC diagnosis by line of therapy | Approximately 2 years
Proportion of patients who receive surgery by stage at treatment | Approximately 2 years
Proportion of patients who receive radiation by stage at treatment | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm